CLINICAL TRIAL: NCT04038918
Title: The Effectiveness of Relaxation Exercises on Pain, Functional Outcomes and Muscle Strength in Patients With Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: The Effectiveness of Progressive Relaxation Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Musa Eymir, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ME-PMR
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Functional Outcomes; Muscle Strength
Keywords: Total knee arthroplasty; progressive muscle relaxation exercise; pain; functional outcomes; muscle strength
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation Exercise Group (Experimental): Standard postoperative physiotherapy program plus progressive muscle relaxation (PMR) exercise will be applied.
  Interventions: Other: progressive muscle relaxation exercise; Other: standard postoperative physiotherapy program
- Control Group (Other): Standard postoperative physiotherapy program will be applied.
  Interventions: Other: standard postoperative physiotherapy program

INTERVENTIONS:
Other: progressive muscle relaxation exercise — In addition to standard postoperative rehabilitation, intervention group will receive PMR exercises focusing on reduce overall body tension, anxiety. The intervention group will perform the PMR exercise in accompanying with a qualified physiotherapist for postoperative 3 days (2 times/day; along 30 minutes for one session).
  Arms: Progressive Muscle Relaxation Exercise Group
Other: standard postoperative physiotherapy program — After surgery, patients will receive standard postoperative rehabilitation program including active-assistive and active range of motion exercises, isometric and isotonic strengthening exercises, gait training and transfer training.

SUMMARY:
The purpose of this study is to investigate the effectiveness of progressive muscle relaxation (PMR) exercise on pain, functional outcomes and muscle strength in patients with TKA. Seventy patients with TKA are going to randomly assigned to intervention group and control group.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is applied in end-stage osteoarthritis to reduce pain, improve functional ability, and provide greater health related quality of life. However, evidence showed that presence of severe pain, impaired functional outcomes and reduced muscle strength continue up to 6 to 12 month after surgery. Relaxation techniques such as progressive muscle relaxation exercise and rhythmic breathing have long been used in treating postoperative pain and for various health-related purposes. Although the number of studies that include relaxation techniques in treating postoperative pain is increasing, there isn't any study that investigate the effectiveness of progressive muscle relaxation exercise on pain, functional outcomes and muscle strength in patients with TKA.

The aim is to investigate the effectiveness of progressive muscle relaxation (PMR) exercise on pain, functional outcomes and muscle strength in patients with TKA.

ELIGIBILITY:
Inclusion Criteria:

* 30 years older above
* Preoperative diagnosis have to be knee osteoarthritis
* Have a primary total knee arthroplasty
* Able to understand Turkish instructions
* Willing and able to attend study

Exclusion Criteria:

* Revision total knee arthroplasty
* Unable to understand verbal and written instructions
* Having previously orthopaedic or neurological disorder that causes gait disturbance

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The Numeric Pain Rating Scale | Postoperative three months
  The Numeric Rating Scale (NPRS), reliable and valid instrument, is commonly used to determine for pain intensity in rehabilitation. The activity and resting pain level in the knee joints will be evaluated by NPRS from 0 to 10 (0 refers to no pain, 10 refers to worst pain).
Iowa Level of Assistance Scale | Postoperative three months
  This test assesses the patient's ability to perform four functional activities, namely, supine to sitting on the edge of the bed, sitting on the edge of the bed to standing, walking 4.57 meters. The scoring of these activities is done as independent 6 points, observational aid 5 points, minimum help 4 points, medium help 3 points, maximum help 2 points, fail 1 point and untested 0 points. Higher values represent a better outcome.
  Speed scoring is done by evaluating the walking speed at a distance of 13.4 meters (44 steps). 20 seconds (sec) and below are recorded as 0, 21-30 sec 1, 31-40 sec 2, 41-50 3, 51-60 sec 4, 61-70 sec 5 and 70 sec. Higher values represent a worse outcome
Hospital for Special Surgery Knee Score | Postoperative three months
  Hospital for Special Surgery knee score. A scoring system evaluation of pain, mobility, range of motion and deforming of the knee giving 0-100 points.
10 meter walk speed test | Postoperative three months
  10MWT testing distance require 5-m acceleration and 5-m deceleration space, with the inner 10-m zone being the distance over which gait is timed. Before the test, patients should be asked to walk as fast as possible and allowed to use assistive devices (cane, walker) if needed. Patients start to walk and accelerate in the 20-m. The stopwatch is started as soon as the patient's leg pass over the starting line and stopped the patient's leg pass over the 10-m sign.
Timed Up and Go (TUG) | Postoperative three months
  To determine fall risk and measure the progress of balance, sit to stand, and walking. The patient starts in a seated position. The patient stands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. The subject is allowed to use an assistive device.
Muscle Strength | Postoperative three months
  Strength of knee muscles will be evaluated by hand-held dynamometer.

SECONDARY OUTCOMES:
Range of Motion | Postoperative three months
  Each patient's active (unassisted) range of knee extension and flexion will be measured, using a goniometer with the patient in the supine position.
The Hospital Anxiety and Depression Scale (HADS) | Postoperative three months
  The HADS aims to measure symptoms of anxiety and depression and consists of 14 items, seven items for the anxiety subscale (HADS Anxiety) and seven for the depression subscale (HADS Depression). Each item is scored on a response-scale with four alternatives ranging between 0 and 3. After adjusting for six items that are reversed scored, all responses are summed to obtain the two subscales. The scoring of HADS is done as normal 0-7 point, borderline case 8-10 points, abnormal case 11-21. Higher values represent a worse outcome.
Tampa Scale for Kinesiophobia (TSK) | Postoperative three months
  The term kinesiophobia refers to a fear of pain with movement - i.e., movements which a patient is hesitant to perform due to fear that the movement will elicit pain. The TSK has been used to assess kinesiophobia in patients with a wide variety of conditions, such as knee disorders. The TSK consists of 17 questions. A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.
12-Item Short Form Survey | Postoperative three months
  SF-12 Health Survey is a shorter version of the SF-36 Health Survey that uses just 12 questions to measure functional health and well-being from the patient's point of view. The SF-12 is a practical, reliable and valid measure of physical and mental health and is particularly useful in large population health surveys or for applications that combine a generic and disease-specific health survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Baker PN, van der Meulen JH, Lewsey J, Gregg PJ; National Joint Registry for England and Wales. The role of pain and function in determining patient satisfaction after total knee replacement. Data from the National Joint Registry for England and Wales. J Bone Joint Surg Br. 2007 Jul;89(7):893-900. doi: 10.1302/0301-620X.89B7.19091. PMID 17673581
- [Background] Bernatzky G, Presch M, Anderson M, Panksepp J. Emotional foundations of music as a non-pharmacological pain management tool in modern medicine. Neurosci Biobehav Rev. 2011 Oct;35(9):1989-99. doi: 10.1016/j.neubiorev.2011.06.005. Epub 2011 Jun 16. PMID 21704068
- [Background] Baird CL, Sands L. A pilot study of the effectiveness of guided imagery with progressive muscle relaxation to reduce chronic pain and mobility difficulties of osteoarthritis. Pain Manag Nurs. 2004 Sep;5(3):97-104. doi: 10.1016/j.pmn.2004.01.003. PMID 15359221